CLINICAL TRIAL: NCT01988181
Title: Blood Volume Monitoring Guided Ultrafiltration Biofeedback on Reduction of Intra-dialytic Hypotensive Episodes in Hemodialysis: A Randomized Cross Over Study
Brief Title: Adjusting Fluid Removal Based on Blood Volume in Hemodialysis: A Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr Jennifer MacRae, Associate Professor Medicine, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BVM-RXOS
Record Dates: First submitted 2013-11-06; First posted 2013-11-20 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Intradialytic Hypotension; End Stage Renal Failure on Dialysis
Keywords: Intradialytic Hypotension; Renal Dialysis; Blood Volume Determination; Clinical Trials, Randomized; Crossover Studies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best clinical practice HD (Active Comparator): All study patients will be dialyzed with the Fresenius 5008 HD machine (Fresenius Medical Care, Bad Homburg, Germany) using high flux dialyzers. For an 8-week period, patients in the best clinical practice (control) phase will use their same prescription as the run-in phase, dialysate sodium of 138mmol/L, dialysate calcium of 1.25mmol/L, dialysate temperature of 36oC, and constant UF rate. BVM will be disabled in this group.
  Interventions: Device: Fresenius 5008 HD machine (Fresenius Medical Care, Bad Homburg, Germany)
- Best clinical practice plus BVM-guided UF biofeedback (Experimental): Patients in the BVM-guided UF biofeedback (intervention) phase will have the same prescription as the control group but will also have the ultrafiltration rate automatically adjusted by the Fresenius 5008 HD machine based on the changes in the relative blood volume.
  Interventions: Device: BVM-UF biofeedback; Device: Fresenius 5008 HD machine (Fresenius Medical Care, Bad Homburg, Germany)

INTERVENTIONS:
Device: BVM-UF biofeedback — The Fresenius 5008 uses an ultrasound and temperature monitor incorporated into the machine to detect ultrasonic velocity and temperature changes to derive the total protein concentration, which is a sum of total plasma proteins and hemoglobin. The relative blood volume is calculated at by dividing the initial concentration of total protein by the total protein concentration at any given time, multiplied by 100. The HD software is based on the critical blood volume entered at the beginning of the dialysis session for each individual patient. The UF rate is adjusted based on the changes in the relative blood volume to the patient's critical relative blood volume.
  Other Names: Fresenius 5008 HD machine with UF control
  Arms: Best clinical practice plus BVM-guided UF biofeedback
Device: Fresenius 5008 HD machine (Fresenius Medical Care, Bad Homburg, Germany) — For an 8-week period, patients in the best clinical practice (control) phase will use their same prescription as the run-in phase, dialysate sodium of 138mmol/L, dialysate calcium of 1.25mmol/L, dialysate temperature of 36oC, and constant UF rate. BVM will be disabled in this group.

SUMMARY:
As kidney function declines, the ability to maintain water balance is impaired and is most often treated with hemodialysis. The removal of excess water in hemodialysis often leads to a sudden drop of blood pressure and causes symptoms of dizziness, light-headedness, cramping, and chest pain. This sudden drop in blood pressure has been linked with complications of heart attacks, strokes and even death. Research has focused on different ways to prevent dangerous drops in blood pressure during hemodialysis. One way is the use of blood volume monitoring biofeedback technology to monitor the patient's relative blood volume and automatically reduce the amount of fluid that is being removed when the blood volume is low to prevent the drop in blood pressure from occurring. This type of biofeedback device is currently available on some hemodialysis machines and while this approach appealing, it is not clear how effective this form of biofeedback is in preventing the drops in blood pressure.

We plan to determine if the use of biofeedback based on the changes in the patient's blood volume will reduce the number of sudden drops in blood pressure that occur during hemodialysis. To do this, we will compare patients treated with this technology to current hemodialysis practices and follow them for important adverse outcomes. The result of interest will be the frequency of hemodialysis sessions complicated by a sudden symptomatic drop in blood pressure. We also plan to monitor the amount of water in the different body compartments, blood pressure, blood pressure medication use, markers of heart function, and patient symptoms and quality of life.

We hope that by providing information on this technology we can reduce the sudden drops in blood pressure in hemodialysis, the associated rates of serious disease or death, and improve patient quality of life.

DETAILED DESCRIPTION:
This is a 22 week parallel group, randomized crossover trial to determine the effect of blood volume monitoring, BVM, guided ultrafiltration (UF) biofeedback on symptomatic intradialytic hypotension (IDH) episodes amongst IDH prone patients. The first part of the study (Part 1 - Run-In/Dialysis Optimization Phase), eligible patients will undergo a four-week run-in phase. During this period all patients will undergo a comprehensive clinical assessment including, clinical weight assessment, anti-hypertensive medication review, and dialysis prescription standardization. At the end of the run-in phase, patients that still meet eligibility criteria will enter the randomized cross-over phase. In part 2 (Randomized Cross-Over Phase), patients are randomized to regular best clinical practice hemodialysis, HD (without BVM-guided UF biofeedback; control arm) or to BVM-guided UF biofeedback (intervention arm) for an 8 week period. This will be followed by a two-week washout phase and then patients will be crossed over for a second 8-week phase. The study will be conducted and reported following the Consolidated Standards of Reporting Trials (CONSORT) 2010 guidelines.

ELIGIBILITY:
Run-in Phase Inclusion Criteria:

* >18 years old
* Maintenance hemodialysis patients for more than 3 months
* Undergo hemodialysis 3-4 times per week for a minimum of three hours per session
* Have >30% of their hemodialysis sessions in the preceding 8 weeks complicated by symptomatic IDH.
* Able to provide written informed consent.

Randomization Phase Inclusion Criteria:

* >18 years old
* Maintenance hemodialysis patients for more than 3 months
* Undergo hemodialysis 3-4 times per week for a minimum of three hours per session
* Have >30% of their hemodialysis sessions in the preceding 4 weeks complicated by symptomatic IDH.

Exclusion Criteria:

* Serum sodium ≤133mmol/L
* Hemoglobin <80g/L
* Active Malignancy
* History of blood transfusions or hospitalizations in the preceding 4 weeks
* Planned change in the renal replacement modality during the planned study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in the rate of symptomatic IDH during hemodialysis | During hemodialysis up to the 22 week study period
  The primary outcome will be rate of symptomatic IDH as defined by an abrupt drop in the systolic blood pressure of ≥20mm Hg when compared to baseline along with an abrupt onset headache, dizziness, unconsciousness, thirst, dyspnea, angina, muscle cramps, or vomiting (reflecting cerebral, cardiac, gastrointestinal, or musculoskeletal ischemia). The end of an episode of IDH will be defined as resolution of the symptom. The number of symptomatic IDH episodes along with the duration of each dialysis treatment will be captured. The rate of IDH for each session will be calculated by dividing the number of episodes by the duration of the session in hours. The rate of IDH will be calculated for every dialysis treatment. The rate of symptomatic IDH will be measured in the two months preceding enrollment, during each phase of the study.

SECONDARY OUTCOMES:
Change in the number of symptomatic IDH per dialysis session | During hemodialysis up to the 22 week study period
  The number of symptomatic IDH episodes in each dialysis treatment will be captured. IDH is defined as in the primary outcome.
Change in the frequency of symptomatic IDH | During hemodialysis up to the 22 week study period
  The number of symptomatic IDH episodes of each dialysis treatment will be captured. IDH is defined as in the primary outcome.
Number and Frequency of Nursing Interventions during hemodialysis | During hemodialysis up to the 22 week study period
  IDH-related nursing interventions are defined as the use of Trendelenburg/supine position, discontinuation of UF, fluid/saline challenge, return of blood, shortened dialysis run, or prolonged (more than 15 minutes) post-dialysis recovery period as a result of IDH or its symptoms. Given the subjective nature of IDH-related symptoms and intervention, in-services and customized dialysis run sheets will be provided to all nurses at participating dialysis centers to ensure that all events are recorded and recorded consistently. The number of symptomatic IDH episodes per session will be record.
Change in Single Session Dialysis Adequacy | After hemodialysis up to the 22 week study period
  Patients that experience symptomatic IDH may require a reduction in the duration of HD treatments with a resultant reduction in dialysis adequacy. Dialysis adequacy will be measured and recorded (usual care) at the end of each dialysis session on the session sheet as single-pooled Kt/V. Single-pooled Kt/v is measured using the previously validated online clearance measurement method, which detects changes in conductivity in the dialysate to reflect the clearance of serum electrolytes and urea.
Electrical Bio-impedance for the determination of change in hydration and fluid status | At the end of the mid-week HD session at week 1, 4, 8, 12, 14, 18, and 22. Up to week 22 study period.
  Whole body and segmental bio-impedance analysis for the determination of fluid composition has been validated in HD patients. Improvement of dry weight has been linked with reduced mortality. Electrical bio-impedance will be performed at the end of the mid-week HD session at week 1, 4, 8, 12, 14, 18, and 22 to determine the total body water, extracellular fluid volume (ECFV), intracellular fluid volume (ICFV), and the ECFV:ICFV ratio.
Change in Serum Brain Natriuretic Peptide (BNP) | At the beginning of the mid-week HD session at week 1, 4, 12, 14, and 22. Up to week 22 study period.
  Chronic hypervolemia in HD is associated with increase in left atrial volume and BNP, which has been shown to predict mortality. Serum BNP will be measured at the beginning of the mid-week HD session at week 1, 4, 12, 14, and 22.
Change in Serum high sensitivity cardiac troponin (hs-Troponin) | At the beginning of the mid-week HD session at week 1, 4, 12, 14, and 22. Up to week 22 study period.
  Biomarkers of cardiac damage such as hs-Troponin are more elevated in HD patients with myocardial stunning and is associated with an increased all-cause mortality. Improved and more frequent dialysis has been associated with a decrease in myocardial stunning, and a trend towards decreasing hs-troponin. Serum hs-Troponin will be performed at the beginning of the mid-week HD session at week 1, 4, 12, 14, and 22.
Change in antihypertensive medication use | At enrollment and the mid-week HD session at week 4, 8, 12, 14, 18, and 22.
  Improvements in a patient's volume status and blood pressure allows for a decrease number or dose of anti-hypertensive medications. The class and number of anti-hypertensive medications will be obtained from the electronic clinical database and subsequently confirmed with a patient interview at enrollment and the mid-week HD session at week 4, 8, 12, 14, 18, and 22. The study investigator will perform medication reconciliation
Relative blood volume Curve | After every hemodialysis session, up to the 22 week study period.
  The shape and slope of the RBV curve has been associated with symptomatic hypotensive episodes in HD. The relative blood volume curve will be downloaded from the Fresenius 5008 dialysis machine to a study computer on a regular basis for all patients in the run-in phase and those in the intervention arm following randomization. The relative blood volume achieved, maximum slope (%/h) of the BVM curve as defined by the percent (%) decline over time (h) will be calculated. The subjective pattern of BVM curve (flat, linear, concave upward, concave downward, regular and irregular line will be determined by the study investigator.
Improvement in Intra-dialytic symptom survey | At the end of each dialysis session, during weeks 1, 4, 8, 12, 14, 18, and 22. Up to the 22 week study period.
  Currently no validated intra-dialytic symptom survey exists to provide an objective measure of intra-dialytic symptom burden. The survey will inquire about the intra-dialytic symptoms of IDH, specifically nausea, vomiting, chest pain, shortness of breath, headache, muscle cramps, dizziness, fainting, fatigue, and anxiety. The survey will be provided by the dialysis nurse, and to be completed by the patient or in conjunction with the dialysis nurse at the end of the dialysis session during weeks 1, 4, 8, 12, 14, 18, and 22. The survey is expected to take less than 1 minute to complete.
Improvement in Inter-dialytic symptom survey | At the beginning of each dialysis session, during weeks 1, 4, 8, 12, 14, 18, and 22. Up to the 22 week study period.
  A survey inquiring about inter-dialytic recovery time to baseline will be provided by the dialysis nurse, and to be completed by the patient or in conjunction with the dialysis nurse at the beginning of dialysis during weeks 1, 4, 8, 12, 14, 18, and 22. The survey will inquire the time it took the patient to recovery from the last dialysis session, is validated in HD patients as a robust assessment quality of life. The survey will take less than 30 seconds to complete.
Assessment of Nursing Perception, Attitudes, and Satisfaction of BVM guided UF biofeedback system | At the end of the control and intervention phase (end of week 12 and 22). Up to the 22 week study period.
  A survey inquiring about nursing perception and attitudes of the BVM guided UF biofeedback will be provided to the nurses at the end of the control and intervention phase. The survey is developed for the purpose of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Quinn, MD PhD, Study Director — University of Calgary; Kelvin Leung, MD, Study Director — University of Calgary; Jennifer MacRae, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Alberta Health Services Southern Alberta Renal Program, Calgary, Alberta, Canada

REFERENCES:
- [Background] Wizemann V, Wabel P, Chamney P, Zaluska W, Moissl U, Rode C, Malecka-Masalska T, Marcelli D. The mortality risk of overhydration in haemodialysis patients. Nephrol Dial Transplant. 2009 May;24(5):1574-9. doi: 10.1093/ndt/gfn707. Epub 2009 Jan 7. PMID 19131355
- [Background] Velasco N, Chamney P, Wabel P, Moissl U, Imtiaz T, Spalding E, McGregor M, Innes A, MacKay I, Patel R, Jardine A. Optimal fluid control can normalize cardiovascular risk markers and limit left ventricular hypertrophy in thrice weekly dialysis patients. Hemodial Int. 2012 Oct;16(4):465-72. doi: 10.1111/j.1542-4758.2012.00689.x. Epub 2012 Apr 20. PMID 22515643
- [Background] Shoji T, Tsubakihara Y, Fujii M, Imai E. Hemodialysis-associated hypotension as an independent risk factor for two-year mortality in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1212-20. doi: 10.1111/j.1523-1755.2004.00812.x. PMID 15327420
- [Background] Selby NM, McIntyre CW. The acute cardiac effects of dialysis. Semin Dial. 2007 May-Jun;20(3):220-8. doi: 10.1111/j.1525-139X.2007.00281.x. PMID 17555488
- [Background] Schreiber MJ Jr. Setting the stage. Am J Kidney Dis. 2001 Oct;38(4 Suppl 4):S1-S10. doi: 10.1053/ajkd.2001.28089. PMID 11602455
- [Background] Schneditz D, Pogglitsch H, Horina J, Binswanger U. A blood protein monitor for the continuous measurement of blood volume changes during hemodialysis. Kidney Int. 1990 Aug;38(2):342-6. doi: 10.1038/ki.1990.207. No abstract available. PMID 2205752
- [Background] Schmidt R, Roeher O, Hickstein H, Korth S. Prevention of haemodialysis-induced hypotension by biofeedback control of ultrafiltration and infusion. Nephrol Dial Transplant. 2001 Mar;16(3):595-603. doi: 10.1093/ndt/16.3.595. PMID 11239038
- [Background] Davenport A. Using dialysis machine technology to reduce intradialytic hypotension. Hemodial Int. 2011 Oct;15 Suppl 1:S37-42. doi: 10.1111/j.1542-4758.2011.00600.x. PMID 22093599
- [Background] Daugirdas JT. Dialysis hypotension: a hemodynamic analysis. Kidney Int. 1991 Feb;39(2):233-46. doi: 10.1038/ki.1991.28. No abstract available. PMID 2002637
- [Background] Dasselaar JJ, Huisman RM, DE Jong PE, Franssen CF. Relative blood volume measurements during hemodialysis: comparisons between three noninvasive devices. Hemodial Int. 2007 Oct;11(4):448-55. doi: 10.1111/j.1542-4758.2007.00216.x. PMID 17922743
- [Background] Agarwal R, Kelley K, Light RP. Diagnostic utility of blood volume monitoring in hemodialysis patients. Am J Kidney Dis. 2008 Feb;51(2):242-54. doi: 10.1053/j.ajkd.2007.10.036. PMID 18215702
- [Background] Agarwal R. Hypervolemia is associated with increased mortality among hemodialysis patients. Hypertension. 2010 Sep;56(3):512-7. doi: 10.1161/HYPERTENSIONAHA.110.154815. Epub 2010 Jul 12. PMID 20625076
- [Derived] Leung KC, Quinn RR, Ravani P, MacRae JM. Ultrafiltration biofeedback guided by blood volume monitoring to reduce intradialytic hypotensive episodes in hemodialysis: study protocol for a randomized controlled trial. Trials. 2014 Dec 10;15:483. doi: 10.1186/1745-6215-15-483. PMID 25496294